CLINICAL TRIAL: NCT05742191
Title: The Effect of Daylight Saving Time Transitions on Sleep and Migraine Headaches.
Acronym: DST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, Sasikanth Gorantla, Neurologist and Sleep Medicine Physician, OSF Healthcare System
Other Study IDs: 1969211
Record Dates: First submitted 2023-02-15; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Episodic Migraine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Established Clinic Patients at OSF INI with Episodic Migraine diagnosis.: Study subjects will be established clinic patients at OSF HealthCare INI neurological institute with a diagnosis of Episodic Migraine.
  Interventions: Other: Daylight Savings time transitions

INTERVENTIONS:
Other: Daylight Savings time transitions — Daylight Savings time transitions.

SUMMARY:
A prospective study that investigates the impact of circadian rhythm disturbances due to daylight saving time transitions on migraine patients.

The Primary aim is to investigate the impact of springtime DST (March 12 2023 at 2 AM on Sunday) on sleep metrics in patients with migraine headaches. Secondary aim is to examine the association between incidence of migraine headaches and sleep metrics with time transitions.

Participants will be provided with a Withings non-wearable/contactless sleep tracker, which will be placed under the mattress for a period of 4 weeks (2 weeks before and 2 weeks after) during daylight saving time transition in March, 2023. Withings Health Mate app will be downloaded to the participant's smartphone to collect Sleep Data. Headache diaries will be provided to log the details of the migraines during the study period. Morningness - eveningness questionnaire (MEQ) will be used to categorize subjects on the chronotype spectrum.

DETAILED DESCRIPTION:
This is a prospective study that investigates the impact of circadian rhythm disturbances due to time transitions on migraine patients. We will seek data analytics assistance to gather the list of subjects who meet the inclusion and exclusion criteria. A thorough review of the electronic medical records will be performed by the PIs to identify the appropriate participants. The Research coordinator will contact the subjects over the phone and discuss the study details. We will follow the numerical order (data as received by the analytics team) and stop contacting the subjects once we reach the target sample size of 50. Interested subjects will be invited to the study visit for formal consenting and the explanation of the study procedure. This study is designed to analyze the sleep metrics (total sleep time, sleep efficiency, sleep onset, and wake up time) in migraine patients with daylight saving spring transition. We will collect the demographics, information regarding migraine headache and Chrono type data to perform required data analysis at OSF HealthCare Illinois Neurological Institute/University of Illinois College of Medicine at Peoria.

Study subjects will be established clinic patients at OSF HealthCare INI neurological institute with a diagnosis of episodic migraines. A total of 50 subjects will be recruited in this study.

Inclusion criteria:

1. Age 18 years and older
2. Episodic migraine diagnosis based on ICHD 3 criteria
3. Subjects with smart phone who can download and use the Health Mate app available on iOS14 and higher and Android 8.0 and higher (Cannot be set up from a computer)
4. Subjects that can commit to sleep on the same bed/mattress every night during the study period
5. Subjects that can commit not to use sleep aids (either prescription or over the counter sleep aids) or sedating medications (sedating anti-depressants, benzodiazepines, anti-histamines, anti-psychotics or gabapentinoids) that assist with sleep onset during the study period.

Exclusion criteria:

1. Patients who do not meet ICHD-3 diagnostic criteria for migraine
2. Patients with migraine diagnosis who are suspected or confirmed to have active medication overuse headaches during the study period.
3. Patients who regularly use sleep aids (either prescription or over the counter sleep aids) or sedating medications (sedating anti-depressants, benzodiazepines, anti-histamines, anti-psychotics or gabapentinoids) to assist with sleep onset.
4. Participants who are planning to initiate new treatment for sleep disorders during the study period.
5. Subjects who participate in shift work.

The PI, Co PI and statisticians shall be the only individuals who will access data. The data will be de-identified at the source and no PHI shall remain connected to any subject's name, date of birth, medical record number, or any other personal information that could tie back to patients once the study is completed.

Withings, under the mattress sleep tracker, will be utilized to collect the sleep metrics in our study https://www.withings.com/us/en/sleep/shop?gclid=CjwKCAjwvNaYBhA3EiwACgndgn_LudRfkDgfsTm9vTfPyIaDs77O7c55PKJa0WZ3W4E0HFqwbIgLhBoCUIwQAvD_BwE&gclsrc=aw.ds

The non-wearable/contactless sleep tracker will be placed under the mattress for a period of 4 weeks (2 weeks before and 2 weeks after) during daylight saving time transition in March, 2023. The device was validated for the detection of sleep apnea; a couple of sleep metrics showed good correlation with the gold standard polysomnogram (PSG) (Total sleep time and sleep efficiency). The Withings sleep tracking mat overestimated TST by 25.8 minutes (PSG - 366.6 (61.2) and Withings device 392.4 (67.2) minutes), acceptable precision. The device estimated sleep efficiency very well when compared to the PSG [PSG - 82.5% and Withings device 82.6%].

The app will be downloaded to the participant's smartphone. The Research Coordinator will contact the subjects who meet inclusion and exclusion criteria to explain the study procedure and obtain informed consent. Subjects will be taught how to download the app and send the data to the study personal at the initial visit. The non-wearable tracking device and the mobile app will be provided free of cost. Mobile app download data includes patient related information (demographics) and sleep metrics. Headache diaries will be provided to log the details of the migraines during the study period. Morningness - eveningness questionnaire (MEQ) will be used to categorize subjects on the chronotype spectrum.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Episodic migraine diagnosis based on ICHD 3 criteria
3. Subjects with smart phone who can download and use the Health Mate app available on iOS14 and higher and Android 8.0 and higher (Cannot be set up from a computer)
4. Subjects that can commit to sleep on the same bed/mattress every night during the study period
5. Subjects that can commit not to use sleep aids (either prescription or over the counter sleep aids) or sedating medications (sedating anti-depressants, benzodiazepines, anti-histamines, anti-psychotics or gabapentinoids) that assist with sleep onset during the study period.

Exclusion Criteria:

1. Patients who do not meet ICHD-3 diagnostic criteria for migraine
2. Patients with migraine diagnosis who are suspected or confirmed to have active medication overuse headaches during the study period.
3. Patients who regularly use sleep aids (either prescription or over the counter sleep aids) or sedating medications (sedating anti-depressants, benzodiazepines, anti-histamines, anti-psychotics or gabapentinoids) to assist with sleep onset.
4. Participants who are planning to initiate new treatment for sleep disorders during the study period.
5. Subjects who participate in shift work.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects will be established clinic patients at OSF HealthCare INI neurological institute with a diagnosis of episodic migraines.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Circadian rhythm disturbances and alteration of total sleep time and sleep efficiency | 4 weeks
  To investigate the impact of springtime DST (March 12 2023 at 2 AM on Sunday) on sleep metrics in patients with migraine headaches.

SECONDARY OUTCOMES:
Migraine Headaches | 4 weeks.
  To examine the association between incidence of migraine headaches and sleep metrics with time transitions.

CONTACTS AND LOCATIONS:
Locations (1):
- OSF HealthCare Saint Francis Medical Center, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mollaoglu M. Trigger factors in migraine patients. J Health Psychol. 2013 Jul;18(7):984-94. doi: 10.1177/1359105312446773. Epub 2012 Oct 26. PMID 23104993
- [Result] Song TJ, Yun CH, Cho SJ, Kim WJ, Yang KI, Chu MK. Short sleep duration and poor sleep quality among migraineurs: A population-based study. Cephalalgia. 2018 Apr;38(5):855-864. doi: 10.1177/0333102417716936. Epub 2017 Jun 22. PMID 28641451
- [Result] Strazisar BG, Strazisar L. Daylight Saving Time: Pros and Cons. Sleep Med Clin. 2021 Sep;16(3):523-531. doi: 10.1016/j.jsmc.2021.05.007. Epub 2021 Jul 2. PMID 34325828
- [Result] Rishi MA, Ahmed O, Barrantes Perez JH, Berneking M, Dombrowsky J, Flynn-Evans EE, Santiago V, Sullivan SS, Upender R, Yuen K, Abbasi-Feinberg F, Aurora RN, Carden KA, Kirsch DB, Kristo DA, Malhotra RK, Martin JL, Olson EJ, Ramar K, Rosen CL, Rowley JA, Shelgikar AV, Gurubhagavatula I. Daylight saving time: an American Academy of Sleep Medicine position statement. J Clin Sleep Med. 2020 Oct 15;16(10):1781-1784. doi: 10.5664/jcsm.8780. PMID 32844740
- [Result] Kantermann T, Juda M, Merrow M, Roenneberg T. The human circadian clock's seasonal adjustment is disrupted by daylight saving time. Curr Biol. 2007 Nov 20;17(22):1996-2000. doi: 10.1016/j.cub.2007.10.025. Epub 2007 Oct 25. PMID 17964164
- [Result] Roenneberg T, Winnebeck EC, Klerman EB. Daylight Saving Time and Artificial Time Zones - A Battle Between Biological and Social Times. Front Physiol. 2019 Aug 7;10:944. doi: 10.3389/fphys.2019.00944. eCollection 2019. PMID 31447685
- [Result] Lahti TA, Leppamaki S, Lonnqvist J, Partonen T. Transition to daylight saving time reduces sleep duration plus sleep efficiency of the deprived sleep. Neurosci Lett. 2006 Oct 9;406(3):174-7. doi: 10.1016/j.neulet.2006.07.024. Epub 2006 Aug 22. PMID 16930838
- [Result] Tyler J, Fang Y, Goldstein C, Forger D, Sen S, Burmeister M. Genomic heterogeneity affects the response to Daylight Saving Time. Sci Rep. 2021 Jul 20;11(1):14792. doi: 10.1038/s41598-021-94459-z. PMID 34285349
- [Result] Sipila JO, Ruuskanen JO, Rautava P, Kyto V. Changes in ischemic stroke occurrence following daylight saving time transitions. Sleep Med. 2016 Nov-Dec;27-28:20-24. doi: 10.1016/j.sleep.2016.10.009. Epub 2016 Nov 2. PMID 27938913
- [Result] Chudow JJ, Dreyfus I, Zaremski L, Mazori AY, Fisher JD, Di Biase L, Romero J, Ferrick KJ, Krumerman A. Changes in atrial fibrillation admissions following daylight saving time transitions. Sleep Med. 2020 May;69:155-158. doi: 10.1016/j.sleep.2020.01.018. Epub 2020 Jan 27. PMID 32088351
- [Result] Prats-Uribe A, Tobias A, Prieto-Alhambra D. Excess Risk of Fatal Road Traffic Accidents on the Day of Daylight Saving Time Change. Epidemiology. 2018 Sep;29(5):e44-e45. doi: 10.1097/EDE.0000000000000865. No abstract available. PMID 29864085
- [Result] Fritz J, VoPham T, Wright KP Jr, Vetter C. A Chronobiological Evaluation of the Acute Effects of Daylight Saving Time on Traffic Accident Risk. Curr Biol. 2020 Feb 24;30(4):729-735.e2. doi: 10.1016/j.cub.2019.12.045. Epub 2020 Jan 30. PMID 32008905
- [Result] Hook J, Smith K, Andrew E, Ball J, Nehme Z. Daylight savings time transitions and risk of out-of-hospital cardiac arrest: An interrupted time series analysis. Resuscitation. 2021 Nov;168:84-90. doi: 10.1016/j.resuscitation.2021.09.021. Epub 2021 Sep 24. PMID 34571135
- [Result] Yadav RK, Kalita J, Misra UK. A study of triggers of migraine in India. Pain Med. 2010 Jan;11(1):44-7. doi: 10.1111/j.1526-4637.2009.00725.x. Epub 2009 Sep 29. PMID 19793343
- [Result] Haque B, Rahman KM, Hoque A, Hasan AT, Chowdhury RN, Khan SU, Alam MB, Habib M, Mohammad QD. Precipitating and relieving factors of migraine versus tension type headache. BMC Neurol. 2012 Aug 25;12:82. doi: 10.1186/1471-2377-12-82. PMID 22920541
- [Result] Negro A, Seidel JL, Houben T, Yu ES, Rosen I, Arreguin AJ, Yalcin N, Shorser-Gentile L, Pearlman L, Sadhegian H, Vetrivelan R, Chamberlin NL, Ayata C, Martelletti P, Moskowitz MA, Eikermann-Haerter K. Acute sleep deprivation enhances susceptibility to the migraine substrate cortical spreading depolarization. J Headache Pain. 2020 Jul 6;21(1):86. doi: 10.1186/s10194-020-01155-w. PMID 32631251
- [Result] Bertisch SM, Li W, Buettner C, Mostofsky E, Rueschman M, Kaplan ER, Fung J, Huntington S, Murphy T, Stead C, Burstein R, Redline S, Mittleman MA. Nightly sleep duration, fragmentation, and quality and daily risk of migraine. Neurology. 2020 Feb 4;94(5):e489-e496. doi: 10.1212/WNL.0000000000008740. Epub 2019 Dec 16. PMID 31843807
- [Result] Smith MT, Edwards RR, McCann UD, Haythornthwaite JA. The effects of sleep deprivation on pain inhibition and spontaneous pain in women. Sleep. 2007 Apr;30(4):494-505. doi: 10.1093/sleep/30.4.494. PMID 17520794
- [Result] Edouard P, Campo D, Bartet P, Yang RY, Bruyneel M, Roisman G, Escourrou P. Validation of the Withings Sleep Analyzer, an under-the-mattress device for the detection of moderate-severe sleep apnea syndrome. J Clin Sleep Med. 2021 Jun 1;17(6):1217-1227. doi: 10.5664/jcsm.9168. PMID 33590821
- [Result] Horne JA, Ostberg O. A self-assessment questionnaire to determine morningness-eveningness in human circadian rhythms. Int J Chronobiol. 1976;4(2):97-110. PMID 1027738